CLINICAL TRIAL: NCT01055418
Title: Cognitive and Cerebral Blood Flow Effects of Vitamin C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, David Kennedy, Professor, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 24AD1
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Endothelial Function; Cognition
Keywords: Vitamin C; Cognitive performance; Cerebral blood flow; Trans cranial doppler; Near infrared spectroscopy
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin C
- Vitamin C (Experimental)
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — Vitamin C will be administered at a dose of 1000mg. There will be at least a 48 hour wash out period between both conditions (placebo and vitamin C), with the order dicteted by Latin square.

SUMMARY:
This investigation is interested in the effects of high dose vitamin C on endothelial function in healthy humans. A high fat meal will be utilized to induce endothelial dysfunction. It is hypothesized that, via antioxidant actions, vitamin C will reverse these effects and in turn improve blood flow- the involvement of nitric oxide suggests that this could extend to cerebral blood flow. This will be monitored by trans cranial doppler flow meter and near infrared spectroscopy.

DETAILED DESCRIPTION:
The acute effect of administering vitamins has received little research attention. The exceptions are a number of studies that have observed that single doses of a variety of vitamins, including Vitamin C, E and several B vitamins, ameliorate endothelial dysfunction in the periphery in participants who smoke, or suffer disorders such as diabetes mellitus and cardio-vascular disease. Endothelial function also varies in healthy people as a consequence of diet, and it is possible that antioxidant vitamins can attenuate the vaso-constriction associated with commonly consumed foodstuffs. Indeed, a study by Title et al (2000) showed that vitamin C improved endothelial function in the forearm following a glucose drink. Given the putative underlying mechanisms involved (e.g. nitric oxide synthesis) any improvement may well also extend to cerebral blood flow (CBF), and therefore improvements in aspects of cognitive function.

The study will therefore assess the effects of a single dose of 1000 mg of vitamin C on cognitive performance and cerebral arterial blood flow velocity (cBFV) using Trans-cranial Doppler, following a high fat meal that has been used in previous endothelial function research.

The high fat meal will be administered 2 hours before testing begins. Research shows that a meal of this type produces effects on the endothelium which are similar to those induced by dysfunctions such as diabetes i.e. blood flow restriction. No adverse effects have been reported with regards this methodology however.

In order to monitor the effects of vitamin C (or not in the case of placebo) on endothelial function and cerebral blood flow near infrared spectroscopy (NIRS) and trans cranial Doppler (TCD) recordings will be taken throughout (in the case of the former technique) and at intermittent stages (in the case of the latter). Both neuroimaging modalities, when used correctly) are entirely safe. Blood pressure readings will also be taken intermittently throughout testing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female,
* 18-35

Exclusion Criteria:

* Smokers,
* not proficient in English,
* are (or are seeking to become) pregnant, are currently taking illicit,
* over the counter/prescription medication (including the contraceptive pill),
* and/or dietary/herbal supplements.
* Food allergies or sensitivities that are relevant to the study,
* a history of/current head trauma,
* learning difficulties,
* ADHD and
* migraines.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Endothelial function (using cerebral blood flow as a proxy measurement as measured by TCD and NIRS. | ~100 mins

SECONDARY OUTCOMES:
Cognitive performance | ~50 mins

CONTACTS AND LOCATIONS:
Overall Officials: David Kennedy, Study Director — Northumbria University
Locations (1):
- Brain, Performance and Nutrition Research Centre, Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom